CLINICAL TRIAL: NCT01172236
Title: Supplementation With Lactoferrin in Preterm Newborns
Acronym: lactoprenew
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Giuseppe Buonocore, Professor, University of Siena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-LF100-2010
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2010-04

CONDITIONS: Prematurity; Low Birth Weight
MeSH Terms: conditions — Premature Birth | interventions — Lactoferrin

ARMS (1):
- Lactoferrin (Experimental)
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin — Experimental group: newborns (group A) will receive a daily dose of 100 mg of lactoferrin (Dicorfam® Elleffe 1''% 2C supplement containing lactoferrin) + standard therapy.
  Control group: newborns (group B) will receive only standard therapy and they will be used as controls.
Drug: Lactoferrin — Experimental group: 650 newborns (group A) will receive a daily dose of 100 mg of lactoferrin (Dicorfam® Elleffe 1''% 2C supplement containing lactoferrin) + standard therapy.Control group: 650 newborns (group B) will receive only standard therapy and they will be used as controls.

SUMMARY:
The main objective of the study is to evaluate the antioxidant effect of lactoferrin and its ability to reduce free radicals related diseases in the newborn. This evaluation will be done through the assessment of neuro-developmental follow-up.

The secondary objective is to identify a panel of markers for assessing oxidative stress and for a correlation with the lactoferrin antioxidant effect.

DETAILED DESCRIPTION:
The study arises from the need to structure care to identify a product natural with antioxidant propriety that may reduce the extent of damage in perinatal neurological disorders related to oxidative stress by limiting the pain for infants and families and simultaneously reducing the cost to the SSN arising from standard pharmacological therapy and rehabilitation in the short and medium term. The research results will remain available to the scientific community and will not be used for profit or commercial. The iron (Fe) is the most abundant transition metal1 in the body and an essential element for growth and welfare of almost all life2 where he played a key role in many biochemical processes3. It is essential as cofactor in many enzymatic reactions and as catalyst in the processes of electron transport, yet is potentially toxic and rarely available. In the presence of oxygen Fe causes harmful action on the cell since it enhances the production by non-enzymatic reactive oxygen species. The hydroxyl radical in particular, can damage various cellular components such as DNA, proteins and membrane lipids. All bodies have therefore developed strategies that allow them to retain Fe was acquired in a soluble, nontoxic and in a form readily available. The Fe excess, also caused by weak bonds that the metal has with nonspecific and specific plasma proteins may carry out its negative effects by generating free radicals through the reactions of Fenton and Heber-Weiss4. Physiological requirements of Fe is higher during periods of rapid growth and differentiation, such as perinatal and nervous system that develops rapidly in late fetal life and early neonatal period, appears to be particularly sensitive to modulations of Fe contents5 In the newborn the inability to regulate, as necessary, the uptake of Fe by the immature gut may be the reason for failure and / or excess metal. Both situations may have adverse effects on neurological development of infants and in case of failure becomes irreversible even6-8 because any supplementation does not improve autcome9-11. In both cases the events that occur in early childhood have adverse effects on neuronal function in adults. The mechanism by which iron deficiency affects brain development is completely unknown but we know that can range up to a general lack metabolic errors of myelination and synaptogenesis and changes in specific funcions12 . It was also suggested that the adverse clinical outcomes in premature infants receiving blood transfusions and / or colonization13 may be related to oxidative damage14-17 <br>The main source of food for newborns is breast milk or formula. Breast milk contains heme Fe consequently the non-heme Fe, which is bound to milk proteins and other substances with lower molecular weight, is the main source of Fe in the diet of infants. The child is able to regulate the absorption of iron from the gut, in response to supplementation, only near the first year of life,18 so the inability of infants to regulate the intestinal absorption predisposes them to a deficiency when the Fe in the diet is insufficient, or an overload, when levels in the diet are high. It was also suggested that the enrichment of Fe in young children may lead to an increase in its plasma concentration and the formation of nonspecific compounds (nonspecific binding to proteins with low affinity bonds) that give rise to the so-called free Fe (NPBI) which originate from reactive oxygen species. Some authors have demonstrated increased oxidative stress in infants of very low birth weight who were subjected to a large oral iron supplementation, especially if breastfed seno.19-21 Although gestational age and some clinical treatments such as transfusions and ventilation considered because of an increased risk of oxidative damage Fe-indotto.22 Since the status of Fe in breast-fed term infants is usually satisfactory, at least until the sixth month, and an important part of Fe in human milk is bound to lactoferrin, has been previously suggested that the effect protective of human milk is related to the presence of this protein fixing most of the Fe and regulates its absorption. The lactoferrin is an iron-binding protein, naturally found in high concentrations in breast milk and in low concentrations in other fluids esocrini23. For the size and structure of lactoferrin is closely linked to another group of Fe-related protein, the transferrin and is considered by many as a member of this family. Lactoferrin binds iron with high affinity binding and its structure is unusually resistant to proteolytic degradation. Besides regulating the absorption of iron during inflammatory processes and infettivi24 performs several physiological functions including antibacterial, antifungal, antivirale25, antiparassitary26, antitumoral27, immunomodulator28-29. This ability antibacterial and antiviral properties, may explain the low prevalence and shorter duration of infection in breast-fed infants. In human milk lactoferrin plays an antioxidant sequestering free ions of Fe30 and thus preventing lipid peroxidation and subsequent milk oxidation31. Some AA.32 have shown this property in vitro using salts and Fe ions in the presence of a biological agent such as reducing ascorbato33. A recent study has also demonstrated its antioxidant effect in blood34. Again lactoferrin is able to bind free Fe, from binding studies, avoiding be sure to trigger a series of chain reactions that produce free radicals and thus reduces the damage induced by oxidative stress. This explains why breastfed children have significantly higher total antioxidant capacity and significantly lower index of oxidative stress. A recent study on infants supplied with formula supplemented with lactoferrin showed that presence of this protein helps the absorption of Fe in the small gut. The same study suggests that its activity could stimulate the proliferation and differentiation of mucosal cells in the gut35, thus increasing the surface and in turn increase the absorption of nutrients. Studies in pregnancy women 36 suggests that lactoferrin may have an anti-inflammatory effect, while also improving the Fe status of women.

ELIGIBILITY:
Inclusion criteria:

* Newborns with a birthweight ≤ 1500 grand/or gestational age ≤ 32 weeks
* Sign of the informed consent by parents

Exclusion criteria:

* Fetal-onset disorders and/or recognizable at birth
* Milk intolerance
* Family history of allergies
* Use of infant formula supplemented with lactoferrin

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1300 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to evaluate the antioxidant effect of lactoferrin and its ability to reduce free radicals related diseases in the newborn. This evaluation will be done trough the assessment of neuro-developmental follow-up. | 12 months

SECONDARY OUTCOMES:
The secondary objective is to identify a panel of markers for assessing oxidative stress and for a correlation with the lactoferrin antioxidant effect. | 24 months